CLINICAL TRIAL: NCT04982640
Title: Establishing Multi-site Feasibility and Fidelity of Yoga to Improve Management of Type-2 Diabetes
Brief Title: Feasibility of Yoga for Type-2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Beth Bock, Ph.D., Senior Research Scientist, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01AT011184
Record Dates: First submitted 2021-07-04; First posted 2021-07-29 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Type2 Diabetes
Keywords: Diabetes; Yoga; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Codes identifying randomization assignment are withheld from the research staff conducting study outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): 12-week program, 60 minutes, twice weekly group-delivered Iyengar yoga
  Interventions: Behavioral: Iyengar yoga; Behavioral: Nutrition Counseling
- Standard Exercise (Active Comparator): 12-week, 60 minutes, twice weekly group-delivered aerobic exercise (e.g., walking) program
  Interventions: Behavioral: Standard Exercise; Behavioral: Nutrition Counseling

INTERVENTIONS:
Behavioral: Iyengar yoga — 60 minute group-classes of Iyengar yoga delivered twice weekly for 12 weeks
  Arms: Yoga
Behavioral: Standard Exercise — 60 minutes, twice weekly for 12 weeks, group-based walking program
  Arms: Standard Exercise
Behavioral: Nutrition Counseling — One, 30-minute session with registered dietitian

SUMMARY:
This study will randomize 90 adults with type-2 diabetes (T2DM) from three different states (RI, MA, and AL) to a 12-week program of either (1) Iyengar yoga or (2) a Standard Exercise program. Follow up assessments occur at 3 and 6-months post-intervention. Results of this study will determine the ability to deliver these interventions with strong rigor and fidelity across multiple sites and will establish the feasibility and acceptability of this intervention across racially and ethnically diverse populations. The study will also examine factors (e.g., outcome expectations, barriers to home practice) that promote long-term adherence to yoga and/or physical activity.

DETAILED DESCRIPTION:
Effective interventions are urgently needed to help adults with Type 2 diabetes (T2DM) achieve and maintain a healthy lifestyle. A significant and growing proportion of Americans, nearly 1 in 10, have T2DM. Uncontrolled diabetes causes serious damage to kidneys, eyes and nerves, and increases risk of heart disease and stroke. Controlling blood glucose is crucial to avoid these complications. Achieving glycemic control requires attention to multiple lifestyle behaviors including healthy eating and regular physical activity. However, only 39 percent of adults with diabetes are physically active. Traditional (western) exercise (e.g., walking and cycling) improves blood glucose levels in adults with T2DM. Long-term adherence is essential to maintain health benefits. However, individuals with T2DM face greater barriers to sustaining physical activity compared to their healthy peers due to the prevalence of overweight and obesity among those with T2DM and the co-morbidities of diabetes (e.g., poor circulation, foot care issues) that create more discomfort during exercise. Yoga is similar to traditional exercise in its ability to improve physical fitness but can be highly accommodating to those with physical limitations. Moreover, as a mindfulness practice, with emphasis on relaxation, meditation, and deep breathing, yoga's effects on stress reduction may have special relevance to people with T2DM. Increased mindfulness leads to improved self-care behaviors including physical activity. Recent meta-analyses suggest a beneficial effect of yoga on glycemic outcomes. However, existing studies have generally been of low quality and conducted with non-US populations.

This U01 application is the next logical step following successful conclusion of our pilot yoga intervention for adults with T2DM (R21AT008830). Feasibility and acceptability were high as measured by program attendance (> 80% of sessions), study completion (92% of participants) and participant satisfaction (M=4.6, +/- 0.57, 1-5 scale). Yoga also improved diabetes selfcare, quality of life and led to reductions in emotional distress and HbA1c. The proposed study will build on these efforts by randomizing a diverse sample of 120 adults with T2DM from three different states (RI, MA, and AL) to a 12-week program of either (1) yoga or (2) Standard Exercise (SE) with follow up at 3 and 6-months post-treatment. Results of this study will determine our ability to deliver these interventions with strong rigor and fidelity across multiple sites and will establish the feasibility and acceptability of this intervention across racially and ethnically diverse populations. We will also examine factors (e.g., outcome expectations, barriers to home practice) that promote long-term adherence to yoga/physical activity. Successful conclusion of this U01 will strengthen future applications for a multi-site RCT to rigorously test the efficacy of yoga for improving HbA1c and diabetes management. If supported, yoga could offer an attractive, sustainable form of physical activity for future diabetes management programs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Diagnosis of type-2 diabetes, stable on medications
3. Physician clearance

Exclusion Criteria:

1. Serious comorbid condition (such as uncontrolled hypertension, glaucoma, heart failure).
2. Complications of diabetes such as diabetic retinopathy, neuropathy and nephropathy
3. Serious psychiatric disorder (e.g. psychosis, major depression, panic attacks, suicidality, or substance dependence).
4. Extremely obese (i.e. Body Mass Index > 45 kg/m2)
5. Currently engaged in yoga, Tai Chi, or other mindfulness-based practice the past six months
6. Pregnant or trying to become pregnant
7. Inability to read and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed as session attendance | 12 weeks
  Each participant is scheduled for 36 classes in total. The percent of classes attended is calculated for each participant to determine feasibility. If the average percentage of classes attended for all participants exceeds 70% the intervention will be deemed feasible.
Acceptability as indicated by participant satisfaction ratings | 12 weeks
  The participant satisfaction scale contains 10 items using a Likert scale from 1 (not at all satisfied) to 5 (very satisfied). Scale items will be summed and averaged for each participant. Scores from all participants are averaged. If the overall average score from all participants is 4 or greater the program will be considered satisfactory.

SECONDARY OUTCOMES:
Hemoglobin A1c | 6 months
  Changes in hemoglobin A1c (HbA1c) from baseline to 6 months follow up
Diabetes Distress as measured by the Problem Areas in Diabetes Scale | 12 weeks
  The problem areas in diabetes scale is a valid and reliable measure of diabetes-related emotional distress. It contains 20 items using a Likert scale from 0 (not a problem) to 4 (serious problem). Scale items are summed and averaged. Higher scores indicate more serious emotional distress associated with managing diabetes.
Fasting Blood Glucose | 12 weeks
  Blood samples taken after > 12 hour fast are assessed using standard laboratory protocols. FBG levels measured as mg/dL at 12 weeks will be compared with baseline values.
Body Mass Index | 6 months
  Measured as body weight in kilograms divided by height in meters squared. [kilograms]/ height [meters2]),

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital- CORO building, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT04982640/ICF_000.pdf